CLINICAL TRIAL: NCT01670747
Title: Evaluation of the Lung Recruitment and End-expiratory Lung Collapse in Patients With Acute Respiratory Distress Syndrome
Brief Title: Evaluation of the Lung Recruitment and End-expiratory Lung Collapse in Acute Respiratory Distress Syndrome (ARDS)
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Other Study IDs: 201208
Record Dates: First submitted 2012-08-14; First posted 2012-08-22 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: ARDS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ARDS: Sedated and mechanically ventilated patients admitted to ICU
  Interventions: Radiation: Chest computed tomography

INTERVENTIONS:
Radiation: Chest computed tomography

SUMMARY:
In this study gas-exchange and respiratory mechanics variations to PEEP change will be correlated to CT lung morphological modifications assessed at different airway pressures (5, 15, 30 and 45 cmH2O).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute lung injury/ acute respiratory distress syndrome
* Mechanical ventilation

Exclusion Criteria:

* Clinical diagnosis of chronic obstructive pulmonary disease
* Clinical diagnosis of pneumothorax
* Haemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to ICU with diagnosis of ARDS who required mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Computer Tomography (CT) scan lung recruitment and CT lung weight | Study day (day 1)
  Aim of the study is to determine the relationship between the opening pressures (recruitment) and closing pressures (PEEP) in order to prevent the opening and closing of the lung parenchyma

CONTACTS AND LOCATIONS:
Overall Officials: Chiumello Davide, MD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

REFERENCES:
- [Background] Gattinoni L, Caironi P, Cressoni M, Chiumello D, Ranieri VM, Quintel M, Russo S, Patroniti N, Cornejo R, Bugedo G. Lung recruitment in patients with the acute respiratory distress syndrome. N Engl J Med. 2006 Apr 27;354(17):1775-86. doi: 10.1056/NEJMoa052052. PMID 16641394
- [Background] Caironi P, Cressoni M, Chiumello D, Ranieri M, Quintel M, Russo SG, Cornejo R, Bugedo G, Carlesso E, Russo R, Caspani L, Gattinoni L. Lung opening and closing during ventilation of acute respiratory distress syndrome. Am J Respir Crit Care Med. 2010 Mar 15;181(6):578-86. doi: 10.1164/rccm.200905-0787OC. Epub 2009 Nov 12. PMID 19910610
- [Derived] Cressoni M, Chiumello D, Algieri I, Brioni M, Chiurazzi C, Colombo A, Colombo A, Crimella F, Guanziroli M, Tomic I, Tonetti T, Luca Vergani G, Carlesso E, Gasparovic V, Gattinoni L. Opening pressures and atelectrauma in acute respiratory distress syndrome. Intensive Care Med. 2017 May;43(5):603-611. doi: 10.1007/s00134-017-4754-8. Epub 2017 Mar 10. PMID 28283699